CLINICAL TRIAL: NCT00004748
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Low-Dose Oral Methotrexate Versus Colchicine for Primary Biliary Cirrhosis
Brief Title: Low-Dose Oral Methotrexate Versus Colchicine for Primary Biliary Cirrhosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Tufts Medical Center (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 199/11664; NEMCH-454
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Liver Cirrhosis, Biliary
Keywords: cirrhosis; gastrointestinal disorders; primary biliary cirrhosis; rare disease
MeSH Terms: conditions — Liver Cirrhosis, Biliary; Fibrosis; Gastrointestinal Diseases; Rare Diseases | interventions — Colchicine; Methotrexate; Ursodeoxycholic Acid

INTERVENTIONS:
Drug: colchicine
Drug: methotrexate
Drug: ursodiol

SUMMARY:
OBJECTIVES:

I. Compare the efficacy of low-dose oral pulse methotrexate (MTX) and ursodiol versus colchicine and ursodiol in patients with primary biliary cirrhosis (PBC).

II. Determine the optimum dose and duration of MTX treatment.

III. Investigate the role of fibrogenic cytokines (FC) in PBC pathogenesis and the effect of treatment on FC production.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

This is a randomized, double-blind study. Patients are stratified by prior/concurrent medical management.

Patients in the first group are treated with oral methotrexate 3 times a week and a daily oral placebo.

Patients in the second group are treated with daily oral colchicine and an oral placebo 3 times a week.

Therapy continues for 10 years. Beginning year 2, daily oral ursodiol is administered to all patients. Patients with disease progression are crossed to the alternate group or undergo liver transplantation if clinically indicated.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Biopsy proven primary biliary cirrhosis (PBC); Disproportionate increase in alkaline phosphatase; Positive antimitochondrial antibody test OR Symptoms consistent with PBC, e.g.: pruritus, fatigue, malaise, jaundice, elevated bilirubin

No clinically advanced PBC, i.e.: bilirubin greater than 10 mg/dL or albumin less than 2.5 g/dL, determined by 2 analyses 10 weeks apart; bleeding esophageal varices or congestive gastropathy; chronic hepatic encephalopathy; chronic ascites

--Prior/Concurrent Therapy-- No concurrent drugs associated with chronic liver disease

--Patient Characteristics--

Hematopoietic: WBC at least 2500 Platelets at least 100,000 (unless due to hypersplenism); Hematocrit at least 30%

Renal: No renal disease that could cause liver dysfunction

Other: No history of alcohol abuse; No other medical illness that might cause liver dysfunction, e.g., severe cardiac failure; No pregnant women

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 1989-11

CONTACTS AND LOCATIONS:
Overall Officials: Marshall M. Kaplan, Study Chair — Tufts Medical Center